CLINICAL TRIAL: NCT03183063
Title: A Novel Method to Detect Pulmonary Thromboembolic Events With Non-Contrast 4DCT
Brief Title: Non-Contrast 4DCT to Detect Pulmonary Thromboembolic Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Guerrero (Other)
Responsible Party: Sponsor-Investigator, Thomas Guerrero, Vice Chair Translational Research, Radiation Oncology, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-018
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Thromboembolisms; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Single Photon Emission Computed Tomography Computed Tomography; Continuous Positive Airway Pressure; Computed Tomography Angiography

STUDY DESIGN:
Intervention Model Description: Patients will be imaged with SPECT/CT and 4DCT to compare perfusion with the respiratory induced blood mass changed (RIBMC) defect. Each patient will have both imaging studies performed on the same day.
  15 subjects will be enrolled into Cohort 1 and will receive SPECT/CT and 4DCT imaging as described. After those are enrolled another 5 subjects will be enrolled into Cohort 2 and will receive SPECT/CT and 4DCT imaging as previously described with the first 4DCT being obtained with normal breathing and the second scan being obtained with positive pressure breathing via BiPAP. Cohort 3 will enroll 124 participants with clinical suspicion of PE, who will be or have had CTA imaging. 4DCT imaging will be performed for these study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 4DCT and SPECT/CT (Experimental): Anticipated 15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. Data will be analyzed for objectives 1, 4 and 5.
  Interventions: Device: 4DCT and SPECT/CT
- 4DCT with BiPAP and SPECT/CT (Experimental): Anticipated 5 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. The second of the two 4DCT scans will be obtained with positive airway breathing via BiPAP. Results in these patients will be analyzed for objective 6 only.
  Interventions: Device: 4DCT with BiPAP and SPECT/CT
- 4DCT with CTA in suspected PE (Experimental): Anticipated 124 participants with CTA ordered/performed for suspected PE will be enrolled to have 4DCT. Goal for analysis is 62 with positive CTA results for PE and 62 with negative CTA results for PE. Data will be analyzed for objectives 2 and 3.
  Interventions: Device: 4DCT with CTA in suspected PE

INTERVENTIONS:
Device: 4DCT and SPECT/CT — Each patient will receive two 4DCT followed by SPECT/CT.
  Arms: 4DCT and SPECT/CT
Device: 4DCT with BiPAP and SPECT/CT — Each patient will receive two 4DCT, with the second scan obtained with positive pressure breathing via BiPAP, followed by SPECT/CT
  Arms: 4DCT with BiPAP and SPECT/CT
Device: 4DCT with CTA in suspected PE — Each patient will receive 4DCT before or after CTA for suspected PE
  Arms: 4DCT with CTA in suspected PE

SUMMARY:
Deep vein thrombosis (DVT) occurs when a blood clot forms in a deep vein, typically in the lower extremities. Pulmonary embolism (PE) occurs when a DVT clot (or fragment) breaks free and travels through the heart to the pulmonary arteries (having to do with the lungs) and lodges in an artery causing a partial or complete blockage. PE is difficult to diagnose due to the non-specific signs and symptoms patients have with this condition such as a cough, shortness of breath, increased heart rate, blood tinged sputum, low oxygen levels.

The standard test to diagnose PE is the Pulmonary Computed Tomography Angiogram (CTA). This can be prohibitive with some patients due to the amount of radiation exposure as well as the complications associated with the need to use intravenous (IV) contrast. In this study the investigators are looking at an alternative method of diagnosing PE's in the Emergency Department where the investigators look at the breathing and blood flow to the lungs thru respiratory gated non-contrast CT (commonly called 4DCT).

The investigators hypothesize that respiratory induced blood mass change in the lungs will allow the identification of under-perfused lung regions.

Cohort 1: An anticipated15 participants will be enrolled with a diagnosis of PE by CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Respiratory induced blood mass change images will be issued from the 4DCT and compared to the SPECT/CT images.

Cohort 2: An anticipated 5 participants will be enrolled under the same criteria and study procedures as Cohort 1. The participants in Cohort 2 will have the addition of Bilevel Positive Airway Pressure (BiPAP) during the 4DCT imaging. This cohort will be used to compare the effect of airway pressure on 4DCT image.

Cohort 3: An anticipated 124 participants will be enrolled. Study procedure will be 4DCT only. Participants must be having or have had a CTA to rule in/out PE. This cohort of the study will be using 4DCT to compare negative CTA to positive CTA findings.

DETAILED DESCRIPTION:
The standard test to diagnose PE is the Pulmonary Computed Tomography Angiogram (CTA). This can be prohibitive with some patients due to the amount of radiation exposure as well as the complications associated with the need to use intravenous (IV) contrast. CTA can detect acute PE with a sensitivity of 99 percent and specificity of 95 percent when combined with CT venography. In patients not medically eligible for CTA, the other option for diagnosis is a ventilation-perfusion (V/Q) single photon emission computed tomography (SPECT) scan. Though this is often prohibitive due to transport to Nuclear Medicine dept., prolonged test time, no test during off hours, etc. In this study the investigators are looking at an alternative method of diagnosing PE's in the Emergency Department where the investigators look at ventilation and perfusion images thru respiratory gated non-contrast CT (commonly called 4DCT).

Technetium-99 m macroaggregated albumin (99mTc-MAA) imaged with single photon emission computed tomography (SPECT) is considered the standard method for the quantitative determination of pulmonary perfusion. Magnetic resonance imaging (MRI) with contrast agents have been utilized experimentally to image the pulmonary vasculature and tissue perfusion. Quantification of SPECT images requires correction of the acquired data for attenuation and attenuation correction, which has lead to the development of SPECT/CT scanners. The low-dose CT can be utilized to evaluate the lung airway architecture, lung parenchyma, and pleural space in conjunction with the registered perfusion images rivaling CTA in sensitivity and specificity.

In a study comparing CT attenuation with SPECT perfusion defects, patients were found to have hypo-attenuated pulmonary regions corresponding to regions with decreased perfusion in 57 percent of acute pulmonary emboli and 88 percent of chronic emboli cases. In the same study, hyper-attenuated regions were found to correspond to regions with hyperperfusion. A method to measure pulmonary perfusion based on subtraction digital fluoroscopy without contrast has been reported. In that study, subtraction images were generated between chest projection images at systole and diastole generating an image representing the perfusion difference. These perfusion projection images were correlate with 99mTc-MAA scintigraphy. Thus, changes in the amount and distribution of pulmonary perfusion throughout the respiratory cycle can be expected and these changes may be apparent on dynamic CT.

Simon described a technique to calculate the change in fractional content of air within pulmonary tissue between anatomically matched CT regions based on a simple model that assumes the density changes were solely due to air content. The investigators successfully applied that model to inhale and exhale breath-hold CT image pairs as well as 4DCT images to create ventilation images. However, the amount of blood in the thorax and lungs varies with the respiratory cycle, thus violating the assumption of this model. The investigators found a cyclic variation in the apparent weight of the lung on 4DCT and others have reported respiratory induced variations in pulmonary perfusion of the lung on MRI. The pulmonary density changes found on 4DCT thus result from both changes in air and blood content.

4DCT derived ventilation images can also be inferred from the respiratory motion induced local tissue volume changes independent of the 4DCT density values. The Jacobian determinant of the deformation field, calculated from the result of images depicting different respiratory phases of the lungs, is used to estimate the local volume changes or ventilation. There is a discrepancy between the density based and the Jacobian based ventilation images suggesting a method to extract respiratory induced blood mass change from 4DCT images. The investigators hypothesize the respiratory induced blood mass changed (RIBMC) will only occur within perfused lung regions. Each image set will contain information representing the density change resulting from both ventilation and RIBMC. Extracting both ventilation and perfusion-like image from the 4DCT image intensities, referred to as Hounsfield Units (HU) is our goal.

The investigators found a cyclic variation in the apparent mass of the pulmonary parenchyma. The investigators hypothesize this variation is due to changes in pulmonary perfusion from respiratory-induced variation in cardiac output. The investigators hypothesize this respiratory induced blood mass change (RIBMC) will allow the identification of hypoperfused lung regions. The investigators did a preliminary study by creating 4DCT RIBMC images from cases with hypoxia induced vasoconstriction, patients with malignant airway constriction. The resulting images compare well with 99mTc-MAA SPECT images. It is unknown, however, if this process works to detect perfusion defects due to PE where the perfusion is obstructed and breathing normal.

In this study patients found to have new segmental, lobar or greater perfusion defects, will be imaged with 99mTc-MAA SPECT/CT and 4DCT to compare perfusion with RIBMC defects. This is a prospective imaging trial of 20 subjects diagnosed by CTA.

An anticipated 15 subjects will be enrolled into Cohort 1 and each will receive 99mTc-MAA SPECT/CT and two (2) 4DCT imaging scans (back-to-back) on the same day. This data will be analyzed for objectives 1, 4 and 5.

An anticipated 5 subjects will be enrolled into Cohort 2 and they will also receive 99mTc-MAA SPECT/CT and two (2) 4DCT imaging scans (back-to-back) on the same day, with the first one being obtained with normal breathing as previously done and the second one being obtained with positive pressure breathing via BiPAP. Cohort 2 results will be analyzed for objective 6 only. Respiratory induced blood mass change (RIBMC) images will be derived from the 4DCT images and quantitatively compared with the SPECT perfusion images.

Cohort 3. The objective of this cohort of the study is to collect and process the image data necessary to assess the sensitivity and specificity of our 4DCT. We will conduct a prospective imaging study of an anticipated 124 patients who present with symptoms leading to a clinical concern for PE and who subsequently undergo chest CTA for further evaluation. One 4DCT before or after the CTA is the only study imaging in this cohort. Data from this cohort will be analyzed for objectives 2 and 3.

Subjects will be followed for a period of 48 hours after imaging for any adverse effects to the 99mTc-MAA.

The Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) will be used to grade all treatment-related adverse events. All Adverse Event (AE) effects will be reported to the Principal Investigator, who will determine the course of action for the study participant and will determine whether the AE affects the study and requires changes to the protocol and/or informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients with segmental or lobar pulmonary emboli on CTA identified within the past 48 hours
* May have initiated anticoagulation therapy
* Patients must sign informed consent to enter this study
* Documented not pregnant if child-bearing age woman

Exclusion Criteria:

* Patients unable to tolerate two 15-minute (4DCT) and one 30-minute imaging sessions (SPECT/CT) in the same day
* Unable to sign informed consent due to cognitive impairment or health status
* Patients who are unstable from a respiratory status requiring ICU care
* Patients who receive tissue plasminogen activator
* Patients who are <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guerrero, MD, PhD, Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Information gathered for this study will not be disclosed to any other person or entity, or for other research.

REFERENCES:
- See also: Abstract on 4DCT ventilation imaging — http://stacks.iop.org/PMB/51/777

RESULTS

PARTICIPANT FLOW:
Groups:
- 4DCT and SPECT/CT: Anticipated15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. Data will be analyzed for objective 1, 4 and 5.
  4DCT and SPECT/CT: Each patient will receive two 4DCT followed by SPECT/CT.
- 4DCT With BiPAP and SPECT/CT: Anticipated 5 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. The second of the two 4DCT scans will be obtained with positive airway breathing via BiPAP. Results in these patients will be analyzed for objective 6 only.
  4DCT with BiPAP and SPECT/CT: Each patient will receive two 4DCT, with the second scan obtained with positive pressure breathing via BiPAP, followed by SPECT/CT. These patients will be analyzed for objective 4 only.
- 4DCT With CTA in Suspected PE: Anticipated 124 participants with CTA ordered/performed for suspected PE will be enrolled to have 4DCT. Goal for analysis is 62 with positive CTA results for PE and 62 with negative CTA results for PE. Data will be analyzed for objectives 2, 3 and 4.
  4DCT with CTA in suspected PE: Each patient will receive 4DCT before or after CTA for suspected PE
Period: Overall Study
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Started | 20 | 4 | 115
Completed | 15 | 0 | 111
Not Completed | 5 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Baseline data included for 15 subjects in Cohort 1, following removal of screen failures and withdrawn subjects. All patients withdrawn from study in Cohort 2, 0 subjects analyzed. 115 subjects included in baseline characteristics for Cohort 3 includes 4 later withdrawn, total 130 subjects.
Groups:
- 4DCT and SPECT/CT: Anticipated15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. Data will be analyzed from this cohort for outcomes 1, 4, and 5.
  4DCT and SPECT/CT: Each patient will receive two 4DCT followed by SPECT/CT.
- 4DCT With BiPAP and SPECT/CT: Anticipated 5 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. The second of the two 4DCT scans will be obtained with positive airway breathing via BiPAP. Data will be analyzed from this cohort for outcome 6 only.
  4DCT with BiPAP and SPECT/CT: Each patient will receive two 4DCT, with the second scan obtained with positive pressure breathing via BiPAP, followed by SPECT/CT. Patients will be compared with Cohort 1 (4DCT and SPECT/CT) for objective 4 only.
- 4DCT With CTA in Suspected PE: Anticipated 124 participants with CTA ordered/performed for suspected PE will be enrolled to have 4DCT. 62 with positive CTA results for PE and 62 with negative CTA results for PE will be included. Data will be analyzed from this cohort for outcomes 2 and 3.
  4DCT with CTA in suspected PE: Each patient will receive 4DCT before or after CTA for suspected PE
- Total: Total of all reporting groups
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE | Total
Number analyzed (Participants) | 15 | 0 | 115 | 130
Age, Continuous [Mean (Full Range); unit: years] | 53.8 [26 to 86] |  | 58.5 [21 to 90] | 57.433 [21 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 64 | 68
  Male | 11 |  | 51 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 |  | 115 | 130

OUTCOME MEASURES:

1. Primary Outcome: Correlation of 4DCT Identified Perfusion With SPECT/CT Identified Perfusion
Description: A custom automated PE detection algorithm will delineate hypo-perfused regions of interest (ROIs) on SPECT perfusion and ROIs on respiratory induced blood mass change (RIBMC) via SPECT/CT. Spatial overlap between hypo-perfused ROIs on SPECT perfusion (standard) and ROIs on RIBMC will be assessed using Dice similarity coefficient (DSC). Spearman correlation will be reported.
Time Frame: 1 hour
Population: Correlation coefficients were only calculated using the 15 subjects with documented PE in Cohort 1 (4DCT and SPECT/CT). All subjects in Cohort 2 (4DCT with BiPAP and SPECT/CT were withdrawn. Subjects in Cohort 3 (4DCT with CTA in suspected PE) were not analyzed for this outcome.
Measure: Median (Full Range); unit: Spearman correlation
Groups:
- 4DCT and SPECT/CT: Anticipated15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. Data will be analyzed for outcomes 1,4 and 5.
  4DCT and SPECT/CT: Each patient will receive two 4DCT followed by SPECT/CT.
- 4DCT With CTA in Suspected PE: Anticipated 124 participants with CTA ordered/performed for suspected PE will be enrolled to have 4DCT. Goal for analysis is 62 with positive CTA results for PE and 62 with negative CTA results for PE. Data will be analyzed for outcomes 2 and 3.
  4DCT with CTA in suspected PE: Each patient will receive 4DCT before or after CTA for suspected PE
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 15 | 0 | 0
Spearman correlation | 0.45 [0.18 to 0.61] |  |

2. Primary Outcome: Count of Participants With True Positive Detection of PE Using Contrast-free 4DCT Functional Imaging and SPECT/CT (Sensitivity)
Description: For each case, an automated PE detection algorithm will determine if functional deficits exist within CT-V and RIBMC. The patient will be classified as PE positive if the algorithm confirms the presence of two or more mismatched segmental or subsegmental defects between CT-V and RIBMC images. This CT-functional imaging (CT-FI) binary classification indicator will be acquired for each patient and compared to the result from the standard acquired CTA. Data will be reported as the count of participants determined to have PE by both imaging modalities (true positives, specificity).
Time Frame: 48 hours
Population: This outcome was analyzed for 51 subjects in Cohort 3 (4DCT with CTA in suspected PE) identified as PE positive by SPECT/CT. All subjects in Cohort 2 (4DCT with BiPAP and SPECT/T) were withdrawn. Subjects in Cohort 1 (4DCT and SPECT/CT) were not analyzed for this objective.
Measure: Count of Participants; unit: Participants
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 0 | 0 | 51
Participants |  |  | 40

3. Primary Outcome: Count of Participants With True Negative Detection of PE Using Contrast-free 4DCT Functional Imaging (Specificity)
Description: For each case, an automated PE detection algorithm will determine if functional deficits exist within CT-V and RIBMC. The patient will be classified as PE negative if the algorithm cannot confirm the presence of two or more mismatched segmental or subsegmental defects between CT-V and RIBMC images. This CT-functional imaging (CT-FI) binary classification indicator will be acquired for each patient and compared to the result from the standard acquired CTA. Data will be reported as count of participants determined not to have PE by both imaging modalities (true negatives, sensitivity).
Time Frame: 48 hours
Population: This outcome was analyzed for 60 subjects in Cohort 3 (4DCT with CTA in suspected PE) identified as PE negative by CTA. All subjects in Cohort 2 (4DCT with BiPAP and SPECT/T) were withdrawn. Subjects in Cohort 1 (4DCT and SPECT/CT) were not analyzed for this objective.
Measure: Count of Participants; unit: Participants
Groups:
- 4DCT and SPECT/CT: Anticipated15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. This data will be analyzed for outcomes 1,4 and 5.
  4DCT and SPECT/CT: Each patient will receive two 4DCT followed by SPECT/CT.
- 4DCT With CTA in Suspected PE: Anticipated 124 participants with CTA ordered/performed for suspected PE will be enrolled to have 4DCT. Goal for analysis is 62 with positive CTA results for PE and 62 with negative CTA results for PE. This data will be analyzed for outcomes 2 and 3.
  4DCT with CTA in suspected PE: Each patient will receive 4DCT before or after CTA for suspected PE
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 0 | 0 | 60
Participants |  |  | 57

4. Secondary Outcome: Measure and Correlate the 4DCT Re-imaging Variance in Radiographic Tidal Volume of RIBMC Images
Description: We will repeat the 4DCT process, obtaining two sets of images, and measure the change in radiographic tidal lung volume on RIBMC between the first and second 4DCT using data from subjects in Cohort 1 (4DCT and SPECT/T). Results are reported as percentage difference between the two scans.
Time Frame: 1 hour
Population: Data was analyzed from the 15 participants in Cohort 1 (4DCT and SPECT/CT). All subjects were withdrawn from Cohort 2 (4DCT with BiPAP and SPECT/CT). Data was not analyzed for this objective for subjects in Cohort 3 (4DCT with CTA in suspected PE).
Measure: Median (Full Range); unit: percentage difference of volume
Groups:
- 4DCT and SPECT/CT: Anticipated15 patients with segmental or lobar pulmonary emboli on CTA. Each will receive SPECT/CT and 4DCT imaging on the same day. Both 4DCT scans will be obtained with normal breathing. Data will be analyzed for objectives 1, 4 and 5.
  4DCT and SPECT/CT: Each patient will receive two 4DCT followed by SPECT/CT.
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 15 | 0 | 0
percentage difference of volume | 14.84 [2.6 to 37.63] |  |

5. Secondary Outcome: Measure and Correlate the 4DCT Re-imaging Variance in Parenchymal Lung Mass of RIBMC Images
Description: We will repeat the 4DCT process, obtaining two sets of images, and measure the change in radiographic parenchymal lung mass on RIBMC between the first and second 4DCT using data from subjects in Cohort 1 (4DCT and SPECT/T). Results are reported as percentage difference between the two scans.
Time Frame: 1 hour
Population: as for outcome 4
Measure: Median (Full Range); unit: percentage difference of mass
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 15 | 0 | 0
percentage difference of mass | 18.23 [0.60 to 38.32] |  |

6. Other Pre Specified Outcome: Measure and Correlate the Airway Pressure Variance of RIBMC Images
Description: An automated PE detection algorithm will detect differences of hypo-perfused regions of interest (ROIs) on 4DCT and deficit ROIs on RIBMC with normal breathing versus positive pressure airway via BiPAP breathing using Dice similarity coefficient (DSC).
Time Frame: 1 hour
Population: Data from cohort 2 (4DCT with BiPAP and SPECT/CT) was to be analyzed for this outcome; however, all subjects were withdrawn. Data is not available from Cohorts 1 (4DCT and SPECT/CT) and 3 ($DCT with CTA in suspected PE) for this outcome measurement.
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | 4DCT and SPECT/CT | 4DCT With BiPAP and SPECT/CT | 4DCT With CTA in Suspected PE
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/4 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/4 | 0/115
Other Adverse Events (participants affected / at risk) | 0/20 | 0/4 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT03183063/Prot_SAP_000.pdf